CLINICAL TRIAL: NCT00860860
Title: Phase I Clinical Study of the Feasibility of Pretargeted Radioimmunotherapy of an Anti-CEA Bispecific Antibody and Lu-177-labeled Peptide in Patients With Advanced Colorectal Cancer
Brief Title: Study of Pretargeted Radioimmunotherapy of a Anti-CEA Bispecific Antibody and Lu177-labeled Peptide in Colorectal Cancer
Acronym: PRIT2008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUNMC-PRIT2008
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Neoplasms
Keywords: radioimmunotherapy; pretargeting; bispecific antibody; lutetium 177; phase I clinical trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Indium-111; Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TF2 — TF2: 75-300 mg
Drug: IMP-288 labeled with In111 and Lu177 — IMP-288: 100 microgram

SUMMARY:
This study will investigate the toxicity, safety and pharmacokinetics of pretargeted radioimmunotherapy with anti-CEA x anti-hapten bispecific antibody TF2 and Lu-177-labeled di-HSG-DOTA peptide IMP-288. Furthermore, the sensitivity of pretargeted imaging with In-111-labeled IMP-288 as compared to standard methods of tumor detection, and the preliminary efficacy of the therapy.

DETAILED DESCRIPTION:
Pretherapy cycle with IMP-288 labeled In111.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CEA expressing advanced colorectal tumors for which no standard treatment is available
* WHO performance status: 0 or 1
* Having normal hematological function: Neutrophils > 1.5 x 109/l; Platelet count > 150 x 109/l, without transfusion during the previous month; Hemoglobin > 5.6 mmol/l
* Total bilirubin < 2 x upper limit of normal (ULN)
* ASAT, ALAT < 3 x ULN
* Serum creatinine < 2 x ULN
* Cockcroft clearance > 50 ml/min
* Negative pregnancy test for women of child¬bearing potential (urine or serum)
* Age over 18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Known metastases to the brain
* Chemotherapy, external beam radiation or immunotherapy within 4 weeks prior to study. Limited field external beam radiotherapy to prevent pathological fractures is allowed, when unirradiated, evaluable lesions elsewhere are present.
* Prior angiogenesis inhibitors within 4 weeks; bevacizumab within 8 weeks
* Cardiac disease with New York Heart Association classification of III or IV
* Patients who are pregnant, nursing or of reproductive potential and are not practicing an effective method of contraception
* Any unrelated illness, e.g. active infection, inflammation, medical condition or laboratory abnormalities, which in the judgement of the investigator will significantly affect patients' clinical status
* Life expectancy shorter than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Toxicity defined by NCI Common Terminology Criteria for Adverse Events version 3.0 | first three weeks: daily, thereafter: weekly

SECONDARY OUTCOMES:
pharmacokinetics and biodistribution of TF2 and Lu-177-labeled IMP-288, sensitivity of pretargeted imaging with In-111-labeled IMP-288, and tumor response using RECIST criteria | Pk/biodistr: first week after administration; imaging: first 5 days after administration of IMP-288-In111; tumor respone: every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: O C Boerman, PhD, Study Chair — RUNMC Department of Nuclear Medicine; R Schoffelen, MD, Study Chair — RUNMC Department of Nuclear Medicine; W JG Oyen, MD PhD, Principal Investigator — RUNMC Department of Nuclear Medicine; W TA van der Graaf, MD PhD, Principal Investigator — RUNMC Department of Medical Oncology
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands